CLINICAL TRIAL: NCT05616000
Title: Comparison of Acetyl- L- Carnitine and Folic Acid Versus Coenzyme Q10 and Folic Acid on Semen and Hormonal Parameters and Semen Oxidative Status in Patients of Primary Infertility. A Double Blind Randomized Clinical Trial
Brief Title: Comparison of Acetyl- L- Carnitine& Folic Acid Versus Coenzyme Q10& Folic Acid on Semen& Hormonal Parameters& Semen Oxidative Status in Patients of Primary Infertility. A Double Blind Randomized Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Mohsin Shah, Associate Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KMU/IBMS/2022/59
Record Dates: First submitted 2022-10-20; First posted 2022-11-14 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Infertility
Keywords: Infertility, Acetyl-L-Carnitine, Coenzyme Q10
MeSH Terms: conditions — Infertility | interventions — Acetylcarnitine; Folic Acid

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetyl-L-Carnitine group (Experimental): Acetyl-L-Carnitine (2gm once a day), folic acid 5mg (once a day) 43 Patients with Primary Infertility will receive Acetyl-L-Carnitine (2gm once a day) orally& folic acid 5mg orally was given to all the participants of this group (once a day).
  Interventions: Drug: Acetyl-l-carnitine, folic acid
- Control group (Experimental): Coenzyme Q10 (400mg once a day) orally was given to all participants& folic acid 5mg (once a day) was also given orally to these participants 43 Patients with Primary Infertility will receive Coenzyme Q10 (400mg once a day), folic acid 5mg (once a day).
  Interventions: Drug: Acetyl-l-carnitine, folic acid

INTERVENTIONS:
Drug: Acetyl-l-carnitine, folic acid — Acetyl-l-carnitine 2gm once a day& folic acid will be given to 43 primary infertile men

SUMMARY:
The investigators aim is to conduct a double blind randomized clinical trial, to study the effects of Acetyl-L-Carnitine and folic acid versus Coenzyme Q10 and folic acid on Semen and hormonal parameters and semen oxidative stress in patients of Primary infertility. Males diagnosed with Primary Infertility are recruited in the study after fulfilling the inclusion nd exclusion criteria. The investigators propose that Primary infertile men may have altered seminal oxidative status & the combinational therapy may achieve favorable seminal , hormonal& antioxidant levels in men having Primary infertility.

DETAILED DESCRIPTION:
Historically, male infertility was considered a taboo subject and its role was deliberately kept in dark until recently when with advances in medical science, the issue was highlighted and its role came into limelight in couple's infertility. Male infertility is mainly caused by oxidative stress. O2- (superoxide anion), OH- (hydroxyl ions), H2O2 (hydrogen peroxide), nitric oxide & ROO- (peroxyl) radicals are all oxygen derived highly reactive oxygen species with a free unpaired electron in their outer orbit making them short lived, highly reactive & unstable. They are produced by the sperms & their normal level help in the sperm maturation, motility, capacitation & facilitation of fertilization. Sperms are at risk of the damage caused by overproduction of these ions. Several factors have been implicated in the overproduction of these reactive oxygen species which include men with testicular hyperthermia (varicocoele, cooks, and drivers) & overproduction by immature sperms & leucocytes. Their overproduction cause damage to the DNA and peroxidation of the lipid membrane leading to detrimental effects on sperms causing infertility There has been no consensus on treatment of male infertility in literature. No standardized treatment is suggested and different treatment combinations are currently been used to manage male infertility. The role of CoQ10 & Acetyl- L-Carnitine is explored recently in the different studies with no consensus on their dosage, duration of treatment & their effect on serum testosterone. This study is conducted to find out the role of Acetyl- L-Carnitine and Co enzyme Q 10 in combination with folic acid and their effect on semen parameters, semen oxidative stress & serum testosterone level in treating primary infertile men.

Objective: To find the effects of Acetyl-l-Carnitine and folic acid versus Coenzyme Q10 and folic acid therapy on sperm parameters, seminal oxidative status & serum testosterone level in primary infertility male patients.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment naïve primary male infertile patients with Oligospermia, Asthenozoospermia , Teratozoospermia & Necrozoospermia
2. Aged between 20 - 45 years
3. Married for more than a year with regular intercourse minimum 3/week.
4. Normal female partner with normal menstrual cycle

Exclusion Criteria:

1. Azoospermic patients
2. Patients with varicocoele
3. Erectile dysfunction
4. Secondary infertility
5. Patients already taking treatment for primary infertility

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2022-08-06 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
change in semen analysis before& after the administration of antioxidants& folic acid. | it will be done at the start of the trial and then after 3 months
  semen analysis of the patients will be done and sperm count million/ml, motility, grading of motility(grade from 0 to 4), volumein ml will be analyzed.
change in seminal oxidative status before& after the administration of antioxidants& folic acid. | it will be done at the start of the trial and then after 3 months
  seminal plasma of the primary infertile men will be analyzed for total antioxidant capacity(TAC)& superoxide dismustase levels through commercially available Elisa kits.
change in serum testosterone in nanograms/dl before& after the administration of antioxidants& folic acid. | it will be done at the start of the trial and then after 3 months
  serum testosterone levels of the patients will be analyzed through commercially available Elisa kits

CONTACTS AND LOCATIONS:
Locations (1):
- Mohsin Shah, PhD, Peshawar, Khyber Pakhtunkha, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wischmann T, Thorn P. (Male) infertility: what does it mean to men? New evidence from quantitative and qualitative studies. Reprod Biomed Online. 2013 Sep;27(3):236-43. doi: 10.1016/j.rbmo.2013.06.002. Epub 2013 Jun 19. PMID 23876974
- [Background] Zegers-Hochschild F, Adamson GD, de Mouzon J, Ishihara O, Mansour R, Nygren K, Sullivan E, van der Poel S; International Committee for Monitoring Assisted Reproductive Technology; World Health Organization. The International Committee for Monitoring Assisted Reproductive Technology (ICMART) and the World Health Organization (WHO) Revised Glossary on ART Terminology, 2009. Hum Reprod. 2009 Nov;24(11):2683-7. doi: 10.1093/humrep/dep343. Epub 2009 Oct 4. PMID 19801627
- [Background] Jarow JP, Sharlip ID, Belker AM, Lipshultz LI, Sigman M, Thomas AJ, Schlegel PN, Howards SS, Nehra A, Damewood MD, Overstreet JW, Sadovsky R; Male Infertility Best Practice Policy Committee of the American Urological Association Inc. Best practice policies for male infertility. J Urol. 2002 May;167(5):2138-44. No abstract available. PMID 11956464
- [Background] Agarwal A, Mulgund A, Hamada A, Chyatte MR. A unique view on male infertility around the globe. Reprod Biol Endocrinol. 2015 Apr 26;13:37. doi: 10.1186/s12958-015-0032-1. PMID 25928197
- [Background] Agarwal A, Saleh RA, Bedaiwy MA. Role of reactive oxygen species in the pathophysiology of human reproduction. Fertil Steril. 2003 Apr;79(4):829-43. doi: 10.1016/s0015-0282(02)04948-8. PMID 12749418
- [Background] Shi JZ, Zhang SS, Zhang Z, Liang Q, Shi Y, Hua JL, Sun T. [Expressions of sperm-specific genes in carnitine-cultured testis sperm of obstructive azoospermia patients]. Zhonghua Nan Ke Xue. 2010 Jun;16(6):504-9. Chinese. PMID 20608353
- [Background] Banihani S, Agarwal A, Sharma R, Bayachou M. Cryoprotective effect of L-carnitine on motility, vitality and DNA oxidation of human spermatozoa. Andrologia. 2014 Aug;46(6):637-41. doi: 10.1111/and.12130. Epub 2013 Jul 3. PMID 23822772
- [Background] Ahmed SD, Karira KA, Jagdesh, Ahsan S. Role of L-carnitine in male infertility. J Pak Med Assoc. 2011 Aug;61(8):732-6. PMID 22355991